CLINICAL TRIAL: NCT06438471
Title: Development of a Novel Soluble Epoxide Hydrolase Inhibitor as a Strategy for Treating Neuropathic Pain in Patients With SCI
Brief Title: Novel Soluble Epoxide Hydrolase Inhibitor for Neuropathic Pain in Patients With Spinal Cord Injury
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: EicOsis Human Health Inc. (Industry)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EC5026-1-04; CDMRP-SC200001 (Other Grant/Funding Number: CDMRP)
Record Dates: First submitted 2024-05-24; First posted 2024-06-03 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Spinal Cord Injuries; Neuropathic Pain
MeSH Terms: conditions — Spinal Cord Injuries; Neuralgia | interventions — EC5026

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EC5026 (Experimental): Multiple oral doses of EC5026
  Interventions: Drug: EC5026 oral tablet
- Placebo (Placebo Comparator): Matching oral placebo
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: EC5026 oral tablet — There will be two ascending dose regimens of EC5026, which will be administered over two consecutive Treatment Periods. During each Treatment Period, EC5026 will be administered orally once daily for 7 consecutive days, with a loading dose on Day 1 and a maintenance dose on Days 2-7 of each treatment period. All study subjects will be enrolled in both Treatment Periods and will receive both dose regimens consecutively, for a total duration of 14 days.
  Oral doses of EC5026 tested in each Treatment Period:
  Treatment Period 1: 6 mg loading dose on Day 1 / 2 mg Maintenance dose on Days 2-7 Treatment Period 2: 8 mg loading dose on Day 8 / 4 mg Maintenance dose on Days 9-14
  Arms: EC5026
Drug: Placebo oral tablet — Participants will be administered a matching oral placebo for 14 consecutive days.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate safety and tolerability of multiple oral doses of EC5026 in male and female patients with neuropathic pain due to spinal cord injury. The main question it aims to answer is whether EC5026 is safe and well tolerated in SCI patients with neuropathic pain. In addition, this trial will also study the effects of EC5026 on pain.

Researchers will compare EC5026 to placebo.

Participants will be asked to:

* Take EC5026 or placebo in a masked fashion, once daily, for 14 consecutive days.
* Undergo physical exams, vital signs assessments, ECGs, and blood draws
* Complete assessments of pain, sleep, functional status, and perception of change

DETAILED DESCRIPTION:
EC5026 has been shown to be effective in preclinical pain models of pain, including inflammatory and neuropathic pain subtypes. Three Phase 1 studies of EC5026 have been conducted in healthy volunteers; a Phase 1a Single Ascending Dose (SAD) study, a Phase 1a Fed-Fasted study, and a Phase 1b Multiple Ascending Dose (MAD) study. The Phase 1b MAD study evaluated the safety, tolerability, and PK of 2 sequential ascending dose regimens of oral EC5026, administered once daily for 7 consecutive days, in healthy volunteers. The present study will evaluate the safety and tolerability, as well as target engagement and pharmacodynamics, of EC5026 administered as multiple doses in subjects with neuropathic pain due to spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet all of the following criteria to be enrolled in this study:

1. Male and female subjects must be 18 and older.
2. Subjects must be willing to provide written informed consent to participate in the study.
3. Subjects must be able to provide own transportation to study site every day for the duration of the study.
4. Subjects must have a complete or incomplete T6-T12 SCI of at least 12 months duration, with below-level neuropathic pain identified by the International Spinal Cord Injury Pain (ISCIP) classification criteria. Importantly, subjects must not be ventilator-dependent as detailed in Exclusion Criteria 1.
5. Subjects must have completed a minimum of 6 of the 7 daily assessments for average and worst daily pain prior to final screening, using an 11-point numerical rating scale (NRS) for average daily pain intensity, and the arithmetic average daily SCI neuropathic pain score must be ≥4 and ≤9, with a standard deviation less than or equal to 1.2. Daily pain assessment screenings will be done over the phone with the study coordinator after informed consent is obtained.
6. Subjects must have failed at least 2 classes of medications for their neuropathic pain due to SCI (classes may include antidepressants, antiepileptics, opioids, anti-inflammatories, topical treatments, etc.).
7. Subjects must be in overall stable condition, as determined by pre-study medical history, physical examination, clinical laboratory tests, and 12 lead ECG measurements
8. Subjects must have normal or not clinically significant clinical laboratory test results, as determined by the study investigator, including coagulation panel, blood cell counts, comprehensive metabolic panel analytes, and creatinine clearance (60 cm3/min or greater). Clinical laboratory tests results that are consistent with known, stable comorbidities will be allowed as long as the comorbidities do not represent an exclusion criteria per se.
9. Subjects must have a negative screening for HIV, Hepatitis C, and Hepatitis B within 30 days of randomization.
10. Subjects must have a normal hypothalamic-pituitary-adrenal and hypothalamic-pituitary-gonadal axes screening study.
11. Subjects must have a negative urinary drug screen (UDS) for illicit drugs (marihuana/THC are allowed) and serum ethanol level <80 mg/dL.
12. Male subjects who are not surgically sterile (vasectomized) and their female sexual partners must agree to use contraception during the study period and for 2 months afterward.
13. Male subjects must not donate sperm during the study and for 12 months after receiving the last dose of study drug.
14. Female subjects must be non-pregnant, non-lactating, and either postmenopausal for at least 1 year, or surgically sterile (bilateral tubal ligation ('clipping or tying tubes' or hysterectomy) for at least 3 months, or they must agree to use two forms of highly effective contraception method (less than 1 pregnancy per 100 people using the method for one year), from 28 days and/or their last confirmed menstrual period prior to study enrollment (whichever is longer) until 2 months after clinic discharge. Postmenopausal status will be defined as follow: minimum 1 year; amenorrhea duration of 12 consecutive months and a serum FSH value >40 IU/L; postmenopausal status must be confirmed by an FSH test at Screening). Highly effective contraception methods include: Intra-uterine device (IUD) containing either copper or levonorgestrel (e.g., Mirena®), and/or barrier methods of contraception, including condoms (external or internal) and diaphragm ('cap'). Hormonal methods of contraception (with the exception of hormonal IUD) are not permitted within this study. Female participants will refrain from using hormonal contraceptives for at least 28 days prior to study entry until the end of the study period. Participants/Participant's partner(s) must also use a barrier form of contraception, from the first dose of study drug through until 2 months after the last dose. For all females of childbearing potential, the pregnancy test result must be negative at Screening and Pre-Study Baseline (Day -1).
15. Subjects must be able to speak, read, and understand English sufficiently to allow comprehension and completion of all study assessments

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from the study:

1. Ventilator-dependent subjects, with the exception of nocturnal use of CPAP or BiPAP.
2. Subjects with pain that is not present every day (chronic) or where the pain description does not have a classic neuropathic phenotype.
3. Subjects with other chronic neuropathic pain conditions, including painful diabetic neuropathy, HIV-associated neuropathic pain, chemotherapy or ethanol-associated neuropathy.
4. Subjects with other pain syndromes that may confound assessment or self-evaluation of the SCI neuropathic pain.
5. Subjects with only negative symptoms, defined as numbness without clear evidence of spontaneous pain, either constant or episodic.
6. Subjects using opioid medications on a regular basis or pro re nata (PRN). Non-opioid pain medications will be allowed if at a fixed stable dose for more than 1 month prior to Screening with no anticipation of the dose changing during the study, and if they do not interfere with the subject's ability to rate pain as per Investigator's discretion. Allowed non-opioid medications include gabapentin, pregabalin, duloxetine, acetaminophen, ibuprofen, celecoxib, meloxicam, other antidepressants including amitriptyline and other antiepileptics, as well as topical capsaicin and topical lidocaine.
7. Subjects with active Hepatitis A, Hepatitis B and/or Hepatitis C.
8. Subjects with any clinically unstable or significant cardiovascular (including acute coronary syndrome within the prior year to Screening), renal, hepatic, respiratory, gastrointestinal, hematological, endocrine, or infectious disease (including HIV infection).
9. Subjects with clinically significant abnormalities on screening vital signs, laboratory tests, and/or ECG. Subjects with poor venous access will also be excluded.
10. Subjects with a history of disorders of the hypothalamic-pituitary-adrenal axis, including adrenal insufficiency and Cushing's, or with a history of disorders of the hypothalamic-pituitary-gonadal axis, including hypogonadism.
11. Subjects who have used any topical, oral, or intravenous exogenous corticosteroids within 12 weeks and/or intra-articular exogenous corticosteroids within 6 months prior to the start of the trial, or who plan on using them during the study.
12. Subjects who have used fludrocortisone or exogenous testosterone products within 12 weeks prior to the start of the trial or who plan on using them during the study.
13. Subjects who have used (within 14 of randomization) or plan on using during the duration of the study any renin-angiotensin system (RAS)-acting drugs (including angiotensin-receptor blockers, or ARBs; angiotensin-converting enzyme inhibitors, or ACE-inhibitors; and direct renin inhibitors) or mineralocorticoid receptor antagonists (such as spironolactone and eplerenone)
14. Subjects who have used chemotherapy agents, or who have a personal history of cancer or cancer in first degree relatives suggestive of elevated cancer risk, other than nonmetastatic skin cancer that has been completely excised, within 5 years prior to Screening.
15. Subjects with a history of bacterial, fungal, or viral infection requiring treatment with antibiotics, antifungal agents, or antivirals within 1 month prior to randomization.
16. Subjects who have used (within 14 days of randomization) or plan on using during the duration of the study any prescription or over-the-counter drugs that are moderate-strong CYP3A4 inducers or inhibitors.
17. Subjects who have used (within 14 days of randomization) or plan on using during the duration of the study any dietary aids, supplements, or foods that are moderate-strong CYP3A4 inhibitors (e.g., grapefruit juice).
18. Subjects with difficulty in swallowing oral medications.
19. Subjects with serious psychosocial comorbidities as determined by the Investigator.
20. Subjects with current cognitive or major psychiatric disorders, or any other condition that could interfere with compliance with study procedures.
21. Subjects with a positive drug or alcohol test (>80 mg/dL) during Screening and/or admission (a positive THC test will be allowed as long as it consists of minimal social use, per discretion of Investigator), or with a recent history of binge drinking within 1 week of randomization.
22. Subjects who have used any other investigational drug within 1 month prior to enrollment. If the investigational drug is known to have a long half-life, a longer washout period will be done.
23. Subjects with a presence or history of active gastrointestinal disorder, including esophageal or gastroduodenal ulceration, or renal, hepatic, or coagulant disorder within 1 month prior to enrollment.
24. Subjects with a family history of significant cardiac disease (i.e., sudden death in first degree relative; myocardial infarction before the age of 50).
25. Subjects with confirmed COVID-19, or suspected COVID-19 (e.g., developed symptoms of a respiratory infection such as cough, sore throat, shortness of breath, or fever, but did not get tested for COVID 19) within 30 days of randomization.
26. Subjects who have received a COVID-19 vaccine within 30 days of randomization or are planning on receiving it during the study duration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAE) [Safety and Tolerability] | 30 days
  All AEs reported or observed during the study will be recorded on the electronic case report forms (eCRF). Information to be collected includes drug treatment, type of event, time of onset, dosage, investigator-specified assessment of severity and relationship to study drug, time of resolution of the event, seriousness, any required treatment or evaluations, and outcome. Any AEs resulting from concurrent illnesses, reactions to concurrent illnesses, reactions to concurrent medications, or progression of disease states must also be reported. All AEs will be followed until they are resolved, stable, or judged by the investigator to be not clinically significant. The Medical Dictionary for Regulatory Activities will be used to code all AEs.

OTHER OUTCOMES:
Effects of 2 ascending multiple dose regimens of EC5026 versus placebo on plasma levels of EC5026 | 30 days
  Standard validated EC5026 measurement platform will be used.
Effects of 2 ascending multiple dose regimens of EC5026 versus placebo on oxylipin biomarkers. | 30 days
  Standard validated oxylipin measurement platform will be used.
Effects of 2 ascending multiple dose regimens of EC5026 versus placebo on target engagement biomarkers. | 30 days
  Target engagement biomarkers will include epoxi fatty acids(EpFA):diol ratio
Effects of 2 ascending multiple dose regimens of EC5026 versus placebo on inflammatory biomarkers: C-Reactive Protein | 30 days
Effects of 2 ascending multiple dose regimens of EC5026 versus placebo on inflammatory biomarkers: IL-6 | 30 days
Effects of 2 ascending multiple dose regimens of EC5026 versus placebo on inflammatory biomarkers: TNF alpha | 30 days
Change in average daily pain from baseline to Day 4 | 4 days
  The average daily pain will be measured as part of the Brief Pain Inventory - Short Form (BPI-SF). This scale uses a 11-point numeric rating scale (NRS) from 0 to 10 to rate pain from "no pain" (score = 0) to "pain as bad as you can imagine" (score = 10).
Change in average daily pain from baseline to Day 8 | 8 days
  The average daily pain will be measured as part of the Brief Pain Inventory - Short Form (BPI-SF). This scale uses a 11-point numeric rating scale (NRS) from 0 to 10 to rate pain from "no pain" (score = 0) to "pain as bad as you can imagine" (score = 10).
Change in average daily pain from baseline to Day 11 | 11 days
  The average daily pain will be measured as part of the Brief Pain Inventory - Short Form (BPI-SF). This scale uses a 11-point numeric rating scale (NRS) from 0 to 10 to rate pain from "no pain" (score = 0) to "pain as bad as you can imagine" (score = 10).
Change in average daily pain from baseline to Day 14 | 14 days
  The average daily pain will be measured as part of the Brief Pain Inventory - Short Form (BPI-SF). This scale uses a 11-point numeric rating scale (NRS) from 0 to 10 to rate pain from "no pain" (score = 0) to "pain as bad as you can imagine" (score = 10).
Change in average daily pain from baseline to Day 21 | 21 days
  The average daily pain will be measured as part of the Brief Pain Inventory - Short Form (BPI-SF). This scale uses a 11-point numeric rating scale (NRS) from 0 to 10 to rate pain from "no pain" (score = 0) to "pain as bad as you can imagine" (score = 10).
Change in average daily pain from baseline to Day 28 | 28 days
  The average daily pain will be measured as part of the Brief Pain Inventory - Short Form (BPI-SF). This scale uses a 11-point numeric rating scale (NRS) from 0 to 10 to rate pain from "no pain" (score = 0) to "pain as bad as you can imagine" (score = 10).
Change in worst daily pain from baseline to Day 4. | 4 days
  The worst daily pain will be measured as part of the Brief Pain Inventory - Short Form (BPI-SF). This scale uses a 11-point numeric rating scale (NRS) from 0 to 10 to rate pain from "no pain" (score = 0) to "pain as bad as you can imagine" (score = 10).
Change in worst daily pain from baseline to Day 8. | 8 days
  The worst daily pain will be measured as part of the Brief Pain Inventory - Short Form (BPI-SF). This scale uses a 11-point numeric rating scale (NRS) from 0 to 10 to rate pain from "no pain" (score = 0) to "pain as bad as you can imagine" (score = 10).
Change in worst daily pain from baseline to Day 11. | 11 days
  The worst daily pain will be measured as part of the Brief Pain Inventory - Short Form (BPI-SF). This scale uses a 11-point numeric rating scale (NRS) from 0 to 10 to rate pain from "no pain" (score = 0) to "pain as bad as you can imagine" (score = 10).
Change in worst daily pain from baseline to Day 14. | 14 days
  The worst daily pain will be measured as part of the Brief Pain Inventory - Short Form (BPI-SF). This scale uses a 11-point numeric rating scale (NRS) from 0 to 10 to rate pain from "no pain" (score = 0) to "pain as bad as you can imagine" (score = 10).
Change in worst daily pain from baseline to Day 21. | 21 days
  The worst daily pain will be measured as part of the Brief Pain Inventory - Short Form (BPI-SF). This scale uses a 11-point numeric rating scale (NRS) from 0 to 10 to rate pain from "no pain" (score = 0) to "pain as bad as you can imagine" (score = 10).
Change in worst daily pain from baseline to Day 28. | 28 days
  The worst daily pain will be measured as part of the Brief Pain Inventory - Short Form (BPI-SF). This scale uses a 11-point numeric rating scale (NRS) from 0 to 10 to rate pain from "no pain" (score = 0) to "pain as bad as you can imagine" (score = 10).
Change in Neuropathic Pain Symptom Inventory (NPSI) total score from baseline to Day 4. | 4 days
  The Neuropathic Pain Symptom Inventory (NPSI) is a questionnaire that assesses neuropathic pain. The total score on the NPSI ranges from 0 to 100, with higher scores indicating more severe pain.
Change in Neuropathic Pain Symptom Inventory (NPSI) total score from baseline to Day 8. | 8 days
  The Neuropathic Pain Symptom Inventory (NPSI) is a questionnaire that assesses neuropathic pain. The total score on the NPSI ranges from 0 to 100, with higher scores indicating more severe pain.
Change in Neuropathic Pain Symptom Inventory (NPSI) total score from baseline to Day 11. | 11 days
  The Neuropathic Pain Symptom Inventory (NPSI) is a questionnaire that assesses neuropathic pain. The total score on the NPSI ranges from 0 to 100, with higher scores indicating more severe pain.
Change in Neuropathic Pain Symptom Inventory (NPSI) total score from baseline to Day 14. | 14 days
  The Neuropathic Pain Symptom Inventory (NPSI) is a questionnaire that assesses neuropathic pain. The total score on the NPSI ranges from 0 to 100, with higher scores indicating more severe pain.
Change in Neuropathic Pain Symptom Inventory (NPSI) total score from baseline to Day 21. | 21 days
  The Neuropathic Pain Symptom Inventory (NPSI) is a questionnaire that assesses neuropathic pain. The total score on the NPSI ranges from 0 to 100, with higher scores indicating more severe pain.
Change in Neuropathic Pain Symptom Inventory (NPSI) total score from baseline to Day 28. | 28 days
  The Neuropathic Pain Symptom Inventory (NPSI) is a questionnaire that assesses neuropathic pain. The total score on the NPSI ranges from 0 to 100, with higher scores indicating more severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: William K Schmidt, PhD, Study Director — EicOsis Human Health Inc.
Locations (1):
- AU Medical Center, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No